CLINICAL TRIAL: NCT05917106
Title: Renal Cancer Monitoring Based on ctDNA Methylomics: A Prospective Cohort Study (MEMORY Study)
Status: Recruiting | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Other Study IDs: 2023DZKY-039-01
Record Dates: First submitted 2023-06-09; First posted 2023-06-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma; Renal Cell Carcinoma; RCC; Kidney Neoplasms; Kidney Cancer
MeSH Terms: conditions — Carcinoma; Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Fresh tumor tissue and blood samplesare collected from each patient.Blood collection time:
  P0: within 7 days before surgery P1:3-7 days after surgery PF1:1 month postoperatively PF2: 4months postoperatively PF3:sequentially 3 months apart PA1: Before postoperative adjuvant therapy PA2: During postoperative adjuvant therapy PA3: After postoperative adjuvant therapy PA4:sequentially spaced 3 months PR: detection when recurrence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To conduct prospective studies to confirm the value of circulating tumor DNA and its abnormal methylation in longitudinal monitoring of patients undergoing kidney cancer surgery.

DETAILED DESCRIPTION:
Some studies have shown the potential of ctDNA in renal cancer monitoring, but the amount of ctDNA released in renal cancer is the lowest among non-cranial tumors. Even in advanced patients, the detection rate of tumor system mutation is less than 50%. DNA methylation is important in the process of tumor occurrence and development. However, no studies have focused on the value of ctDNA methylation in monitoring renal cancer, nor have large prospective cohort studies been conducted in patients with renal cancer.

This study intended to analyze the dynamic changes of circulating tumor DNA and its methylation status in patients with kidney cancer from preoperative to long-term follow-up, and to compare the evaluation value of methylation detection with traditional imaging examination and traditional blood tumor markers in the monitoring process.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed renal cell carcinoma
* Without any treatment
* Agree and accept radical surgical treatment
* Signed written informed consent
* ECOG(Eastern Cooperative Oncology Group) performance is 0 or 1
* Follow up protocol and related procedures

Exclusion Criteria:

* Had other cancers
* Had received any antitumor therapy before
* Known or suspected active autoimmune disease
* Informed consent is not possible due to medical or psychiatric problems
* Have clinical symptoms or diseases of the heart that are not well controlled
* Patients judged by the investigators to be unsuitable for inclusion in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RCC patients undergoing surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
To explore the predictive effect of ctDNA methylomics on the prognosis and medication guidance of renal carcinoma. | 5 years
To explore the advance time of ctDNA methylomics in monitoring postoperative recurrence of renal cancer compared with imaging. | 5 years
The molecular mechanism of renal cancer recurrence was analyzed with baseline tissue and circulating methylation profiles. | 5 years
A renal cancer recurrence risk model was established based on clinical information, molecular risk factors and ctDNA methylomics | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, China, Nanjing, Jiangsu, China